CLINICAL TRIAL: NCT03049800
Title: Is Cognitive Training Neuroprotective in Early Psychosis?
Status: Completed | Type: Observational
Sponsor: University of Minnesota (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Other Study IDs: PSYCH-2017-25501; R21MH110208-01A1 (NIH)
Record Dates: First submitted 2017-01-26; First posted 2017-02-10 (Actual); Last update posted 2021-02-16 (Actual); Status verified 2021-02

CONDITIONS: Psychosis; Healthy
Keywords: Recent onset psychotic illness; Healthy controls; Cognitive training; 7T Magnetic Resonance Imaging; Prisma 3T Magnetic Resonance Imaging
MeSH Terms: conditions — Psychotic Disorders | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (4):
- FEP - Treatment as Usual: First Episode Psychosis patients who receive treatment as usual while participating in an associated randomized controlled trial examining the effect of computerized cognitive training.
  Interventions: Device: Magnetic Resonance Imaging
- FEP - Targeted Cognitive Training: First Episode Psychosis patients who receive targeted cognitive training exercises while participating in an associated randomized controlled trial examining the effect of computerized cognitive training.
  Interventions: Device: Magnetic Resonance Imaging
- FEP - General Cognitive Exercises: First Episode Psychosis patients who receive general cognitive exercises while participating in an associated randomized controlled trial examining the effect of computerized cognitive training.
  Interventions: Device: Magnetic Resonance Imaging
- Healthy Controls: Age and gender matched controls who are psychologically and physically healthy will be recruited from the community to participate in this cohort.
  Interventions: Device: Magnetic Resonance Imaging

INTERVENTIONS:
Device: Magnetic Resonance Imaging — Functional, structural, and diffusion weighted imaging conducted with a 7T-PS scanner and a Prisma 3T scanner.

SUMMARY:
The purpose of this study is to perform longitudinal high-resolution 7T MRI and Prisma 3T MRI in participants with first-episode psychosis (FEP) enrolled in our ongoing randomized controlled clinical trial (RCT) of cognitive training. The investigators seek to determine whether a 12-week course of intensive cognitive training of auditory processing in young FEP patients delivered remotely as a stand-alone treatment is neuroprotective against neural tissue loss in auditory cortex (superior temporal gyrus, STG), and possibly in other cortical regions. The investigators will also observe the effects of training on white matter integrity in the brain.

DETAILED DESCRIPTION:
The current protocol seeks to examine whether cognitive training can prevent accelerated gray matter loss and promote changes in the functional connectome in first-episode psychosis patients. Specifically, we aim to use Prisma 3T and 7T imaging to examine functional, structural, and diffusion weighted images to determine whether these treatments can influence neural plasticity. Scanning will be done at the Center for Magnetic Resonance Research (CMRR) at the University of Minnesota. Participants will complete three approximately one-hour scanning sessions on the 3T Siemens Prisma scanner and three approximately one-hour scanning sessions on the 7T-AS scanner. We aim to use scan sequences compatible with the Human Connectome Project both for purposes of cross collaboration and data sharing.

This study will seek to enroll 80 participants. 60 participants will be considered First Episode Psychosis (FEP) patients, meaning that they have been diagnosed with a psychotic illness and have started receiving treatment at a First Episode Psychosis clinic (following the NAVIGATE model) within the last two years prior to enrollment. These participants will be recruited from a separate study protocol conducted by Dr. Sophia Vinogradov which examines remote cognitive training in FEP subjects (Minnesota Community-Based Cognitive Training in Early Psychosis, NCT03079024). 20 of these participants will receive treatment as usual (TAU), 20 will be assigned to Targeted Cognitive Training (TCT), and 20 will be assigned to Generalized Cognitive Exercises (GCE). Additionally, the investigators will enroll 20 healthy, age and gender matched controls (HC). All participants will undergo one 7T MRI and one Prisma scan at three time points: Baseline; Post-Intervention/12-weeks; and 6 month follow up.

The three 3T scan sessions will be matched as closely as possible, given hardware limitations, to the HCP 3T imaging protocol described here: http://protocols.humanconnectome.org/HCP/3T/imaging-protocols.html. This will include ~16 minutes of 3D structural imaging using MP-RAGE and T2-weighted scans, ~14 minutes of resting state fMRI relying on a gradient-echo EPI sequence, and 18 minutes of diffusion weighted MRI relying on a spin-echo EPI sequence. Scan parameters for acquisitions will seek to match the HCP Lifespan data acquired to date on the CMRR Prisma 3T.

For 7T scans, we will collect a standard T1-weighted MP2-RAGE structural scan, 12 minutes of resting fMRI using standard gradient-echo EPI sequences, and a diffusion-weighted DTI sequence compatible both with HCP and 7T-AS hardware. To maximize use of high-resolution imaging techniques while balancing ease of access and use, we aim to use the Siemens 7T-AS scanner with the NOVA 32-Channel head coil optimized for both structural and functional imaging.

Specific Aims

1. Use the Siemens Prisma 3T MRI system and 7T MRIs to investigate longitudinal changes in brain gray matter volume in left Heschl gyrus (HG) and left planum temporale (PT) between baseline, post-training (approximately 12 weeks), and 12 months, within 20 FEP subjects who have undergone targeted cognitive training of auditory processing and 20 FEP subjects who have undergone general cognitive exercises, as compared to 20 treatment-as-usual FEP subjects and 20 age and gender matched healthy controls. Secondarily, we will also examine gray matter volume changes in prefrontal, parietal, and left hippocampual cortex.
2. Use the Siemens Prisma 3T MRI system and 7T MRI to investigate longitudinal changes in left temporal lobe white matter integrity between baseline, post-training (approximately 12 weeks), and 12 months, within 20 FEP subjects who have undergone targeted cognitive training of auditory processing and 20 FEP subjects who have undergone general cognitive exercises, as compared to 20 treatment-as-usual FEP subjects and 20 age and gender matched healthy controls. Secondarily, we will also examine changes in left superior longitudinal fasiculus, left arcuate fasciculus, left uncinated fasciculus, left uncinated fasciculus, cingulum bundle, and corpus callosum.
3. Investigate the association of changes in brain gray matter volume and white matter integrity with changes in clinical, cognitive and functional outcome measures in the FEP subjects who have undergone training.

Exploratory Aims

1. Use Prisma 3T and 7T MRI to explore longitudinal changes between baseline, post-training (approximately 12 weeks), and at 6 month follow-up, in a novel putative MRI diffusion imaging biomarker that may represent neuroinflammation (extracellular volume fraction) in 20 FEP subjects who have undergone targeted cognitive training and 20 FEP subjects who have undergone general cognitive exercises, as compared to 20 treatment-as-usual FEP subjects and 20 age and gender matched healthy controls.
2. Investigate the association of these changes with clinical, cognitive, and functional outcomes in the subject groups.

ELIGIBILITY:
First Episode Psychosis (FEP) Participants

Inclusion Criteria:

* Enrolled in the Mini-COTES randomized controlled trial examining cognitive training in First Episode Psychosis (NCT03079024)
* Clinical diagnosis of schizophrenia, schizoaffective disorder, schizophreniform disorder, major depressive disorder with psychotic features, bipolar disorder with psychotic features, psychosis disorder not otherwise specified, or unspecified schizophrenia spectrum disorder, and started receiving treatment services at a First Episode Psychosis Program within the last two years
* Good general physical health
* Age between 16 and 35 (inclusive)
* Fluent in written and spoken English
* No neurological disorder (diagnosis of Autism Spectrum Disorder is allowed)
* Achieved clinical stability, defined as outpatient status for at least one month prior to study participation, stable doses of psychiatric medications for at least one month prior to study participation
* Women who are pregnant or breastfeeding may participate in this study

Healthy Controls (HC) Participants

Inclusion Criteria:

* Age between 16 and 35 (inclusive)
* Fluent in English
* Good general physical health
* No neurological disorder
* No current or past diagnosis of a psychotic disorder, mood disorder, or anxiety disorder

All Participants

Exclusion Criteria:

* Unable to provide informed consent (or assent if under 18)
* Parents do not provide consent for participants under 18
* Clinically significant substance abuse that is impeding the subject's ability to participate fully during recruitment, assessment, or training (is unable to remain sober for assessments).
* Cannot pass the CMRR safety screen for receiving an MRI
* Participant does not comply with study procedures. Exclusion is determined at PI discretion.

Ages: 16 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: FEP participants will be currently enrolled in "Minnesota Community Based Cognitive Training in Early Schizophrenia," NCT03079024. This study examines cognitive training delivered remotely to patients who receive treatment for FEP at a NAVIGATE-model clinic. There are three groups in this study: one receives targeted cognitive training (TCT); one receives general cognitive exercises (GCE); and the third receives treatment-as-usual (TAU). Cognitive training groups complete up to 30 hours of training over 6-12 weeks. 20 participants in each arm will be recruited for a total of 60.
  Control subjects who are matched to the FEP participants in age and gender will be recruited from the community. We will recruit a total of 20 psychologically and physically healthy adults for this study.
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2017-06-12 (Actual); Primary Completion 2021-02-15 (Actual); Study Completion 2021-02-15 (Actual)

PRIMARY OUTCOMES:
Longitudinal changes in gray matter volume | 1 year
  The investigators will conduct 3 7T and 3 Prisma 3T structural and functional MRI scans over a period of 10-12 months to observe any changes in gray matter volume between cohorts and over time. The investigators will examine gray matter volume in the left Heschl gyrus (HS), left planum temporale (PT), and the prefrontal, parietal, and hippocampal cortices.
Longitudinal changes in white matter integrity | 1 year
  The investigators will conduct 3 7T and 3 Prisma 3T diffusion weighted MRI scans over a period of 10-12 months to observe any changes in white matter integrity between cohorts and over time. The investigators will examine changes in the left temporal lobe, left superior longitudinal fasiculus, left arcuate fasciculus, left uncinated fasciculus, left uncinated fasciculus, cingulum bundle, and corpus callosum.
Association of changes in gray matter volume and white matter integrity with changes in clinical, cognitive and functional outcome measures in FEP participants | 1 year
  The investigators will compare the longitudinal changes in gray matter volume and in white matter integrity to the changes in measures of clinical, cognitive, and functional assessments in the associated randomized controlled study of cognitive training (NCT03079024), between cohorts and over time. The investigators will examine the differences between participants who received cognitive training and those who received treatment as usual.

SECONDARY OUTCOMES:
Longitudinal changes in extracellular volume fraction | 1 year
  The investigators will examine changes in MRI diffusion imaging of this novel biomarker that may represent neuroinflammation. The investigators will examine the changes between cohorts and over time.
Association between longitudinal changes in extracellular volume fraction and changes in clinical, cognitive, and functional outcomes in FEP participants. | 1 year
  The investigators will compare the longitudinal changes in extracellular volume fraction to the changes in measures of clinical, cognitive, and functional assessments in the associated randomized controlled study of cognitive training (NCT03079024), between cohorts and over time. The investigators will examine the differences between participants who received cognitive training and those who received treatment as usual.

CONTACTS AND LOCATIONS:
Overall Officials: Sophia Vinogradov, MD, Principal Investigator — University of Minnesota Department of Psychiatry
Locations (1):
- University of Minnesota, Dept of Psychiatry, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Yes
Data from this study will be shared with the NIMH Data Archive, ID C2788. Additionally, interested collaborators may reach out to the PI directly to share data.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Supporting information will be made available one year after completion of all study procedures, and will be available indefinitely.
Access Criteria: Interested researchers may access this data using the NIMH Data Archive by following the requirements of this registry. Those who would like to see other supporting information may reach out to the PI directly. The PI may share data at their discretion, according to institutional policies, which may include entering into a Data Use Agreement and accessing data within a data shelter.